# STATISTICAL ANALYSIS PLAN (SAP)

Protocol Number: GEN-003-005

Protocol Title: A Randomized, Placebo-controlled, Double-blind

Study to Assess the Efficacy and Safety of a Maintenance Dose of GEN-003 in Subjects with

Genital Herpes Infection

Product Name or Number: GEN-003

Sponsor: Genocea Biosciences, Inc.

Cambridge Discovery Park 100 Acorn Park Drive, 5<sup>th</sup> Floor

Cambridge, MA 02140

SAP Prepared by:

Thomas H. Oliphant, PhD

Andrew Kampfschulte, MS

Biostatistician

Innovative Analytics, Inc. 161 East Michigan Ave. Kalamazoo, MI 49007

USA

SAP Version Number (Date): Version 1.0 (February 7, 2018)

# TABLE OF CONTENTS

| 1 | I | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 4 |
|---|-----|------------------------------------------------|----|
| 2 | S | STUDY OVERVIEW | 5 |
| 3 | 5 | STUDY OBJECTIVES | 6 |
| | 3.1 | Primary Efficacy Objective | 6 |
| | 3.2 | Secondary Efficacy Objectives | 6 |
| | 3.3 | Safety Objective | 6 |
| 4 | A | ANALYSIS POPULATIONS | 6 |
| | 4.1 | Modified Intent-to-Treat Population | 6 |
| | 4.2 | Safety Population | 6 |
| | 4.3 | Per Protocol Population | 6 |
| 5 | S | STATISTICAL METHODOLOGY | .7 |
| | 5.1 | Summarization of Data | 7 |
| | 5.2 | Sample Size Justification | 7 |
| | 5.3 | Randomization | 7 |
| | 5.4 | Unblinding | .7 |
| | 5.4 | .1 At Subject Level | .7 |
| | 5.4 | 2 Interim Analysis | .7 |
| | 5.4 | 3 Final Analysis | .7 |
| | 5.5 | Data Handling | 8 |
| | 5.5 | .1 Method for Handling Missing Data | 8 |
| | 5.5 | 2 Definition of Baseline Values | 8 |
| | 5.5 | .3 Windowing of Visits | 8 |
| | 5.5 | .4 Justification of Pooling | 8 |
| | 5.5 | .5 Withdrawals, Dropouts, Loss to Follow-up | .8 |
| | 5.6 | Output Production and Validation | 8 |
| 6 | 5 | SUBJECT DISPOSITION | 8 |
| 7 | I | DEMOGRAPHIC CHARACTERISTICS | .9 |
| 8 | N | MEDICAL HISTORY | 9 |
| Q | ( | CONCOMITANT MEDICATIONS | 0 |

| 10 | ELECTRONIC DIARY COMPLIANCE | 9 |
|---|---|---|
| 11 | EFFICACY ANALYSIS | 9 |
| 11. | .1 Genital Herpes Lesion Rate | 9 |
| 11. | 2 Frequency of Genital Herpes Recurrences | 10 |
| 11. | 3 Proportion of Subjects Recurrence-Free | 10 |
| 11. | .4 Time to First Genital Herpes Recurrence | 10 |
| 11. | .5 Duration of Genital Herpes Recurrences | 10 |
| 11. | .6 Antiviral Medication Use | 10 |
| 12 | SAFETY ANALYSES | 11 |
| 12. | .1 Reactogenicity | 11 |
| 12. | 2 Adverse Events | 11 |
| 13 | SUBJECT LISTINGS | 11 |
| 14 | INTERIM ANALYSIS | 11 |
| 15 | FINAL SIGN-OFF FOR Genocea Biosciences, Inc Protocol GEN-003-005<br>STATISTICAL ANALYSIS PLAN | 12 |
| 16 | REVISIONS TO STATISTICAL ANALYSIS PLAN | 13 |
| 17 | APPENDIX | 14 |
| 17. | .1 Conventions for Statistical Tables and Listings | 14 |

# 1 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation or Term | Definition |
|----------------------|----------------------------------------------|
| AE | adverse event |
| AESI | adverse event of special interest |
| DMC | Data Monitoring Committee |
| EQ-5D-5L | EuroQol – 5 Domains – 5 Levels |
| IA | interim analysis |
| IM | intramuscular |
| MAAE | medically attended adverse event |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified intent-to-treat |
| MM2 | Matrix-M2 adjuvant |
| PP | Per protocol |
| PT | Preferred term |
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | standard deviation |
| SOC | System Organ Class |

#### 2 STUDY OVERVIEW

This study is a randomized, double-blind, placebo-controlled clinical trial of GEN-003 in subjects who have received previous doses of GEN-003. Subjects who completed Study GEN-003-003 and received all 3 doses, reported data in daily electronic reporting period on at least 80% of days, and had no important protocol deviation in that trial were offered enrollment in this study. Subjects who met all inclusion and no exclusion criteria and provided written informed consent for this study were randomized within 11 to 18 months after the last active GEN-003 dose in a 1:1 ratio to receive 1 intramuscular (IM) dose (the maintenance dose) of GEN-003 or placebo. Randomization was stratified on the basis of the GEN-003 dose received by the subject in Study GEN-003-003.

Subjects were to use a daily electronic tool for reporting the presence or absence of genital herpes lesions and severity of genital herpes symptoms from Day 1 until the Month 6 visit.

Subjects were to complete the EuroQol -5 Domains -5 Levels (EQ-5D-5L) questionnaire on each day of the first recurrence after the maintenance dose through Month 6.

Local reactions and systemic events were to be recorded for the first 7 days after the maintenance dose on a paper Diary Card; if any event was ongoing after Day 8, it was to be followed until resolution. All adverse events (AEs) and concomitant medications were to be recorded from Day 1 to Day 29/Month 1. After Day 29/Month 1 to the end of the study, only serious AEs (SAEs), AEs of special interest (AESIs), medically attended AEs (MAAEs), antiviral medications, and vaccines were to be recorded. All AEs were to be graded in accordance with the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials from Grade 1 (mild) to Grade 4 (life-threatening).

From Month 2 to Month 6, the investigational site was to contact each subject monthly by telephone or site visit for review of daily electronic reporting tool data and assessment of SAEs, AESIs, and antiviral medication use (through Month 6).

A Data Monitoring Committee (DMC) was to review safety data at intervals of a minimum of 3 months until all subjects have completed the GEN-003/placebo dosing period. Any additional meetings and the specific safety monitoring plan were to be detailed in the DMC charter.

#### 3 STUDY OBJECTIVES

## 3.1 Primary Efficacy Objective

The primary efficacy objective is as follows:

• To evaluate the efficacy of GEN-003 versus placebo administered as a maintenance dose in reduction of genital herpes lesion rate

# 3.2 Secondary Efficacy Objectives

The secondary efficacy objectives are as follows:

- To evaluate the efficacy of GEN-003 versus placebo administered as a maintenance dose on genital herpes recurrence through Month 6:
- Reduction of genital herpes recurrence frequency
- Increase of proportion of subjects who are genital herpes recurrence-free
- Increase of time to first genital herpes recurrence
- Reduction of genital herpes recurrence duration

# 3.3 Safety Objective

• To evaluate the safety and tolerability of a maintenance dose of GEN-003 versus placebo

#### 4 ANALYSIS POPULATIONS

# 4.1 Modified Intent-to-Treat Population

The Modified Intent-to-Treat (mITT) population includes all randomized subjects who received the maintenance dose. Subjects will be analyzed according to the treatment to which they were randomized.

# 4.2 Safety Population

The Safety population includes all randomized subjects who received the maintenance dose. Subjects will be analyzed according to the treatment received.

# 4.3 Per Protocol Population

The Per Protocol (PP) population includes subjects who received the maintenance dose, reported data during the daily electronic reporting period on at least 80% of days, and had no important protocol deviations. Subjects will be analyzed according to the treatment received.

#### 5 STATISTICAL METHODOLOGY

#### 5.1 Summarization of Data

Study results will be summarized in tabular format by treatment group (GEN-003, Placebo), with descriptive statistics and/or in subject listings. In general, descriptive statistics for continuous variables will consist of subject count, mean, standard deviation (SD), median, and range; and descriptive statistics for categorical variables will consist of subject counts and percentages. Time-to-event data will be analyzed by the Kaplan-Meier life test method, and results will be summarized by 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals (CIs), as well as the percentage of censored observations.

The efficacy analyses described in this Statistical Analysis Plan (SAP) will be performed for the mITT and PP populations. The safety analyses will be performed for the safety population.

## **5.2 Sample Size Justification**

Sample size in this study is dependent on the enrollment in GEN-003-003. No formal sample size calculations were performed for this study.

#### 5.3 Randomization

Eligible subjects were randomized in a 1:1 ratio to receive 1 IM dose of GEN-003 (60  $\mu$ g each antigen and 50  $\mu$ g MM2) or placebo. Randomization was stratified on the basis of the GEN-003 dose received by the subject in Study GEN-003-003.

# 5.4 Unblinding

#### 5.4.1 At Subject Level

Unblinding of treatment assignment is discouraged. If a medical emergency occurrs for which the identity of the treatment assignment is critical to the care of a subject, the Investigator will call the Medical Monitor to discuss. If unblinding is deemed necessary, a designated unblinded study team member (unblinded statistician) will provide the treatment assignment to the Medical Monitor who will provide the information to the Investigator.

#### 5.4.2 Interim Analysis

The Sponsor and members of the study team will be unblinded to the treatment arms at the interim analysis time point. Only the DMC members and unblinded statistician will have access to unblinded safety data at the subject level and only at specified intervals throughout the study or as necessary to perform the task of overall safety monitoring.

#### 5.4.3 Final Analysis

After database lock at the end of the study, individual subject treatment assignments will be unblinded and available to all study team personnel, including the lead, blinded statistician.

## 5.5 Data Handling

#### 5.5.1 Method for Handling Missing Data

No imputation of missing data will be performed. All available safety and efficacy data will be included in data listings and summaries.

#### **5.5.2** Definition of Baseline Values

Unless otherwise specified, Baseline values are defined as the values collected on Day 1 of GEN-003-005.

## 5.5.3 Windowing of Visits

All data will be categorized based on the scheduled visit at which it was collected. These visit designators are predefined values that appear as part of the visit tab in the electronic case report form.

#### 5.5.4 Justification of Pooling

All data from all sites will be pooled. Study center or treatment-by-center interaction will generally not be included in statistical analyses.

## 5.5.5 Withdrawals, Dropouts, Loss to Follow-up

Time-to-event variables will be censored if a subject withdraws, drops out, or is lost to follow-up before the documentation of the time to the first subject-reported recurrence after the maintenance dose.

If a subject withdraws, drops out, or is lost to follow-up before the first recurrence after the maintenance dose is recorded, the subject will be censored at the last documented time without recurrence recorded; if no record is available after the maintenance dose, the subject will be censored at Day 1.

# 5.6 Output Production and Validation

All analyses will be performed using SAS V 9.2 or higher (SAS Institute, Inc, Cary, North Carolina, USA). Validation and quality control of the tables, listings, and figures that display the results of the statistical analysis of the data from this study will follow the appropriate Innovative Analytics standard operating procedures.

#### 6 SUBJECT DISPOSITION

A breakdown of the number and percentage of subjects enrolled by site and treatment group will be provided. The number of subjects who complete the study will be summarized in tabular format for the safety population. Reasons for discontinuation from the study will also be summarized. A summary of analysis populations table by treatment group will be presented, and a subject listing of protocol deviations will be produced.

#### 7 DEMOGRAPHIC CHARACTERISTICS

Demographic and baseline characteristics will be summarized by treatment group.

For quantitative variables, summary statistics (number [n], mean, SD, minimum, median, and maximum) will be presented for all subjects. For qualitative variables, results will be summarized as counts and percentages for all subjects.

## 8 MEDICAL HISTORY

All medical history events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system. Medical history events (past and current medical disorders) will be presented by treatment group for the safety population, summarized by MedDRA system organ class (SOC) and preferred term (PT).

## 9 CONCOMITANT MEDICATIONS

All medications will be coded using the World Health Organization (WHO) Drug Dictionary. Frequency tables will be presented by treatment group that summarize the prior and concomitant medications taken during the course of the study. A subject listing of medications will also be provided.

#### 10 ELECTRONIC DIARY COMPLIANCE

Summary statistics will be presented by treatment group for the electronic diary compliance after the maintenance dose.

#### 11 EFFICACY ANALYSIS

# 11.1 Genital Herpes Lesion Rate

Lesion rate (days) is defined as number of days with lesions divided by the time period of follow-up for lesions (in days). The days with lesions will be collected continuously throughout the study via an electronic lesion diary, and lesion rates will be calculated for the following periods: Baseline and Day 1 to 183 (post-dosing). For the purposes of determining days with lesions, a diary entry of missing will be treated the same as a diary entry of "no," except in the following case: if 1 or 2 consecutive instances of missing is flanked by "yes" values on both sides, those missing values will be treated as a "yes" value.

Lesion rate will be analyzed with descriptive summary tables for overall and individual lesion rates calculated for the periods noted above. Individual subject lesion rates will be compared for the active treatment group vs. placebo using the Wilcoxon rank sum test.

## 11.2 Frequency of Genital Herpes Recurrences

The frequency of genital herpes recurrences in the 6-month period after the maintenance dose will be calculated as the number of recurrences reported using the daily electronic lesion diary, and will be summarized by mean, SD, median, and range. The median frequencies of recurrences will be compared between treatment groups using the Wilcoxon rank sum test.

## 11.3 Proportion of Subjects Recurrence-Free

The proportion of subjects in each treatment group who are genital herpes recurrence-free at 6 months after the maintenance dose will be tabulated and compared using a chi-square test for homogeneity of proportions.

## 11.4 Time to First Genital Herpes Recurrence

Time to the first subject-reported recurrence in the 6 month period after the maintenance dose will be estimated via Kaplan-Meier approach. The log rank test will be used to compare time to first recurrence between the GEN-003 and placebo arms.

## 11.5 Duration of Genital Herpes Recurrences

Mean lesion outbreak duration is defined as the average number of days with lesions per outbreak for those who have lesion outbreaks (recurrences).

Mean lesion outbreak duration will be presented in a similar descriptive summary table as done for lesion rate as described above. Individual subject mean outbreak duration will be summarized by treatment arm over 6 months (Days 1 to 183) after the maintenance dose. A Wilcoxon rank sum test will be used to test the hypothesis that the median mean lesion outbreak durations are the same between treatment groups at 6 months after the maintenance dose.

#### 11.6 Antiviral Medication Use

Antiviral medications will be coded using the most current WHO Drug Dictionary and summarized by anatomical therapeutic chemical class and preferred term with results presented by treatment group. Antiviral medication use (Y/N) during the 6 months following the maintenance dose will be summarized by treatment group.

#### 12 SAFETY ANALYSES

# 12.1 Reactogenicity

Frequency counts will be presented for systemic events and local reactions for the safety population. This will be done for events occurring within the first 7 days following the maintenance dose. Results will be presented by treatment group and maximum severity. Duration, in days, of events will also be summarized with n, median, minimum and maximum. All analyses will be done for the safety population.

Antipyretic and analgesic medications taken within 7 days after the maintenance dose will also be summarized by treatment group.

#### 12.2 Adverse Events

All AEs will be coded using the MedDRA coding system. Frequency tables will be presented by treatment group for all AEs by SOC and PT. Frequency tables will be produced for AEs leading to discontinuation of dosing, by severity, by causality, for most common (≥5% in any group) AEs, SAEs, MAAEs, and AESIs. Subject listings of all AEs by study day will also be provided.

In all displays, AEs will be displayed by MedDRA SOC and PT, with subjects who have the same AE counted only once for that event and with subjects who have more than 1 AE within a SOC counted only once in that SOC.

#### 13 SUBJECT LISTINGS

All data that are collected and entered into the study database will be presented in subject listings by GEN-003-005 treatment group.

#### 14 INTERIM ANALYSIS

An interim analysis (IA) will be conducted after all subjects should have completed the Month 6 visit and will include analysis of lesion rates. The tables to be produced for this interim analysis are noted in the List of Statistical Tables Table of Contents (TOC) with an 'X' in the IA column.

# 15 FINAL SIGN-OFF FOR GENOCEA BIOSCIENCES, INC PROTOCOL GEN-003-005 STATISTICAL ANALYSIS PLAN

| Thomas H Oliphant Thomas H Oliphant (Feb 22, 2018) | Feb 22, 2018 |
|---|---|
| Thomas H. Oliphant, PhD<br>Biostatistician<br>Innovative Analytics | Date |
| • MD (Feb 22, 2018) | Feb 22, 2018 |
| Seth Hetherington, M.D.<br>Chief Medical Officer<br>Genocea Biosciences, Inc. | Date |
| <u>Tingting Ge</u> Tingting Ge (Peb 22, 2018) | Feb 22, 2018 |
| Tingting Ge, PhD Director of Biostatistics Genocea Biosciences, Inc. | Date |

CONFIDENTIAL 12

# 16 REVISIONS TO STATISTICAL ANALYSIS PLAN

| Date | Revision | Statistician's Signature |
|------|----------|--------------------------|
| • | • | • |
| • | • | • |
| • | • | • |
| • | • | • |
| • | • | • |
| • | • | • |

## 17 APPENDIX

## 17.1 Conventions for Statistical Tables and Listings

The following conventions are used in the mockups for the statistical tables:

[Sponsor] = [Genocea Biosciences]

[Protocol] = [GEN-003-005]

[Drug name] = [GEN-003]

In general, font size will be Courier 9-point and all margins will be 1 inch.

**Treatment Groups** 

GEN-003 Antigens  $60 \mu g / M2 50 \mu g$ 

Placebo

## **List of Statistical Tables for GEN-003-005**

| Table No. | Table Title | Analysis<br>Population | IA |
|---|---|---|---|
| 14.1.1 | Number and Percentage of Enrolled Subjects by Site and Treatment Group | Safety | |
| 14.1.2 | Demographic and Baseline Characteristics by Treatment Group | Safety | X |
| 14.1.3 | Summary of Analysis Populations by Treatment Group | | |
| 14.1.4 | Subject Disposition by Treatment Group | Safety | |
| 14.1.5 | Frequency of Medical History Events by Treatment Group | Safety | |
| 14.1.6 | Prior Medications by Treatment Group | Safety | |
| 14.1.7 | Concomitant Medications by Treatment Group | Safety | |
| 14.1.8 | Summary of Antiviral Medications Taken During the Study by Treatment Group, Drug Class and Preferred Term | Safety | |
| 14.2.1 | Summary Statistics for Electronic Diary Compliance After Maintenance Dose by Treatment Group | mITT | |
| 14.2.2.1 | Descriptive Summary of Overall Lesion Rates by Treatment Group and Observation Period | mITT | X |
| 14.2.2.2 | Descriptive Summary of Overall Lesion Rates by Treatment Group and Observation Period | PP | |
| 14.2.3.1 | Descriptive Summary of Individual Subject Lesion Rates by Treatment Group and Observation Period | mITT | X |
| 14.2.3.2 | Descriptive Summary of Individual Subject Lesion Rates by Treatment Group and Observation Period | PP | |

| Table No. | Table Title | Analysis<br>Population | IA |
|---|---|---|---|
| 14.2.4.1 | Frequency of Recurrences at 6 Months After Maintenance Dose by Treatment Group | mITT | X |
| 14.2.4.2 | Frequency of Recurrences at 6 Months After Maintenance Dose by Treatment Group | PP | |
| | | | 1 |
| 14.2.5.1 | Proportion of Subjects Who Are Recurrence Free at 6 Months After Maintenance Dose | mITT | X |
| 14.2.5.2 | Proportion of Subjects Who Are Recurrence Free at 6 Months After Maintenance Dose | PP | |
| 14.2.6.1 | Time to First Recurrence After Maintenance Dose | mITT | X |
| 4.2.6.2 | Time to First Recurrence After Maintenance Dose | PP | |
| 14.2.7.1 | Descriptive Summary and Analysis of Mean Lesion Outbreak Duration Over 6 Months After Maintenance Dose | mITT | X |
| 14.2.7.2 | Descriptive Summary and Analysis of Mean Lesion Outbreak Duration Over 6 Months After Maintenance Dose | PP | |
| 14.2.8.1 | Summary of Antiviral Medication Use After Maintenance Dose | mITT | |
| 14.2.8.2 | Summary of Antiviral Medication Use After Maintenance Dose | PP | |
| 14.3.1.1 | Frequency Table of All Adverse Events by SOC, Preferred Term, and Treatment | Safety | |
| 14.3.1.2 | Frequency Table of All Adverse Events by SOC, Preferred Term, Treatment, and Severity | Safety | |
| | Trequency 1 and 011 m 1 av or 02 Events of 000, 11010 man, 110 and 10110, and 00 vortey | Saroty | |

| Table No. | Table Title | Analysis<br>Population | IA |
|---|---|---|---|
| 14.3.1.4 | Frequency Table of All Adverse Events Leading to Discontinuation of Dosing by SOC, Preferred Term and Treatment | Safety | |
| 14.3.1.5 | Frequency Table of Subjects with Adverse Events of Special Interest by SOC, Preferred Term, and Treatment | Safety | |
| 14.3.1.6 | Frequency Table of All Adverse Events with ≥ 5% Occurrence by SOC, Preferred Term, and Treatment | Safety | |
| 14.3.1.7 | Summary of Local Reactions and Systemic Events Occurring Within 7 Days Postdose by Treatment and Maximum Severity | Safety | |
| 14.3.1.8 | Descriptive Summary of Duration (days) of Systemic Events and Local Reactions by Treatment | Safety | |
| 14.3.1.9 | Summary of Antipyretic/Analgesic Medications Taken Within 7 Days after Maintenance Dose by Treatment Group, Drug Class, and Preferred Term | Safety | |
| 14.3.2.1 | Frequency Table of Subjects with Serious Adverse Events by SOC, Preferred Term, and Treatment | Safety | |
| 14.3.2.2 | Frequency Table of Subjects with Medically Attended Adverse Events by SOC, Preferred Term, and Treatment | Safety | |

Protocol: [Protocol number] page x of y

Number and Percentage of Enrolled Subjects by Site and Treatment Group Table 14.1.1:

Safety Population

| | sarety ropurat | 1011 |
|-----------|------------------------------------|-----------------|
| Site | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
| Site 1 | n (x.x%) | n (x.x%) |
| Site 2 | n (x.x%) | n (x.x%) |
| Site 3 | n (x.x%) | n (x.x%) |
| Site 4 | n (x.x%) | n (x.x%) |
| etc. | | |
| Site X | n (x.x%) | n (x.x%) |
| All Sites | n (x.x%) | n (x.x%) |

Date Produced: mm/dd/yy Program:

Demographic and Baseline Characteristics by Treatment Group Table 14.1.2: Safety Population

| Saf | ety Population | | |
|------------------------|----------------|----------|------------|
| | GEN-003 60 ug/ | | |
| | M2 50 ug | Placebo | Total |
| | N=xx | N=xx | N=xx |
| Variable | | | |
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Sex | | | |
| Male | n (x.x%) | n (x.x%) | n (x.x%) |
| Female | n (x.x%) | n (x.x%) | n (x.x%) |
| Race | | | |
| American Indian or | n (x.x%) | n (x.x%) | n (x.x%) |
| Alaska Native | | | |
| Asian | n (x.x%) | n (x.x%) | n (x.x%) |
| Black | n (x.x%) | n (x.x%) | n (x.x%) |
| Hawaiian or Pacific | n (x.x%) | n (x.x%) | n (x.x%) |
| Islander | | | |
| White | n (x.x%) | n (x.x%) | n (x.x%) |
| Other | n (x.x%) | n (x.x%) | n (x.x%) |
| Ethnicity | | | |
| Hispanic or Latino | n (x.x%) | n (x.x%) | n (x.x%) |
| Not Hispanic or Latino | n (x.x%) | n (x.x%) | n (x.x%) |
| Weight (lbs) | | | |
| n | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | xx.xxx | XX.XXX |
| Median | XX.XX | xx.xx | XX.XX |
| Min, Max | XX.X, XX.X | xx.x, | XX.X, XX.X |
| | , | xx.x | • |

Program:

Date Produced: mm/dd/yy

[Sponsor]

Protocol: [Protocol number] page x of y

Table 14.1.3: Summary of Analysis Populations by Treatment Group

| Population | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
|---|---|---|
| Modified Intent-to-Treat[a] | n (x.x%) | n (x.x%) |
| Safety[b] | n (x.x%) | n (x.x%) |
| Per Protocol[c] | n (x.x%) | n (x.x%) |

[a] Includes all randomized subjects who received the maintenance dose.

[b] Includes all randomized subjects who received the maintenance dose.

Program: Date Produced: mm/dd/yy

<sup>[</sup>c] Includes all subjects in the mITT Population who reported 80% of daily electronic reporting data, and who had no major protocol deviations

Protocol: [Protocol number] page x of y

Table 14.1.4: Subject Disposition by Treatment Group

Safety Population GEN-003 60 ug/ M2 50 ug Placebo Disposition N=xxN=xxSubject completed the study n (x.x%) n (x.x%) Primary Reason for Discontinuation from Study Withdrew consent for reason other than AE n (x.x%)n (x.x%) Withdrew consent due to solicited or unsolicited AEs Lost to Follow-up n (x.x%) n (x.x%) Non-compliance n (x.x%) n (x.x%) Investigator discretion n (x.x%) n (x.x%) Sponsor request n (x.x%) n (x.x%) Death n (x.x%) n (x.x%)

n (x.x%)

n (x.x%)

n (x.x%)

n (x.x%)

Program: Date Produced: mm/dd/yy

Site termination

Study termination

Protocol: [Protocol number] page x of y

Table 14.1.5: Frequency of Medical History Events by Treatment Group

Safety Population

| Salety Pop | Julation | | |
|---|---|---|---|
| Medical History Events | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx | |
| SOC1 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event1 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event2 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event3 | n (x.x%) | n (x.x%) | |
| SOC2 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event4 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event5 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event6 | n (x.x%) | n (x.x%) | |
| | n (x.x%) | n (x.x%) | |
| SOC3 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event7 | n (x.x%) | n (x.x%) | |
| Preferred Term for MH Event8 | n (x.x%) | n (x.x%) | |
| ETC | | | |
| | | Dat | e Produced: |

Program:

Programming Notes:

• Data comes from Medical History module

- Sort by SOC and preferred terms
- These data will be coded in MedDRA.

Protocol: [Protocol number] page x of y

Table 14.1.6: Prior Medications by Treatment Group

Safety Population

| | оритистоп | |
|---|---|---|
| ATC Text Level 2<br>Preferred Name | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
| AMO Mont Torrel 2 | . ( ) | ( % ) |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |

Date Produced: mm/dd/yy

Note: Prior Medication mapping was based on WHODRUG.

Program:

Programming Note:

• Prior medications are those medications with a start date BEFORE date of maintenance dose (Day 1).

Protocol: [Protocol number] page x of y

Table 14.1.7: Concomitant Medications by Treatment Group

Safety Population

| Salety ropulation | | |
|---|---|---|
| ATC Text Level 2<br>Preferred Name | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |
| ATC Text Level 2 | n (x.x%) | n (x.x%) |
| Preferred Name1 | n (x.x%) | n (x.x%) |
| Preferred Name2 | n (x.x%) | n (x.x%) |
| Preferred Name3 | n (x.x%) | n (x.x%) |

Note: Concomitant Medication mapping was based on WHODRUG.

Program:

Programming Note:

• Concomitant medications are those medications with a start date on or after date of maintenance dose (Day 1), or with a start date before Day 1 and continue beyond Day 1.

Date Produced: mm/dd/yy

Protocol: [Protocol number] page x of y

Table 14.1.8: Summary of Antiviral Medications Taken During the Study by Treatment Group, Drug Class and Preferred
Term

Safety Population Day 1 to Month 6

| Preferred Term | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
|---|---|---|
| Any Antiviral Medication | n (x.x%) | n (x.x%) |
| Preferred Term 1 | n (x.x%) | n (x.x%) |
| Preferred Term 2 | n (x.x%) | n (x.x%) |
| Preferred Term 3 | n (x.x%) | n (x.x%) |
| etc. | | |

Program: Date Produced: mm/dd/yy

#### Programming Notes:

• Antiviral medications are defined as medications with an ATC2 Class of 'ANTIVIRALS FOR SYSTEMIC USE'

Protocol: [Protocol number] page x of y

Table 14.2.1: Summary Statistics for Electronic Diary Compliance After Maintenance Dose by Treatment Group

| mITT Popula | ation | |
|--------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=XX |
| Days with Entry | | |
| n | XX | XX |
| Mean | xx.xx | XX.XX |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| | xx.x, xx.x | xx.x, |
| Min, Max | | XX.X |
| Days without Entry | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| | xx.x, xx.x | XX.X, |
| Min, Max | | XX.X |
| Percent Compliance | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | xx.xxx | XX.XXX |
| Median | xx.xx | XX.XX |
| | xx.x, xx.x | xx.x, |
| Min, Max | | XX.X |

Note: Days with Entry are days from Day 1 to Month 6 visit or date of discontinuation with an entry of 'Yes' or 'No' Days without Entry are days from Day 1 to Month 6 visit or date of discontinuation with an entry of blank

Program: Date Produced: mm/dd/yy

Programming Notes:

- Use Day 1 as start date
- Use earliest of Month 6 visit and date of completion or early termination (dsdtdat) from Subject Disposition form as cutoff date
- Percent Compliance = Days with Entry/(Days with Entry + Days without Entry) \* 100%

Protocol: [Protocol number] page x of y

Table 14.2.2.1: Descriptive Summary of Overall Lesion Rates by Treatment Group and Observation Period

mITT Population Variable Visit GEN-003 60 ug/ Statistic M2 50 ug Placebo N=xxN=xxOverall lesion rate (days) Days with lesions/followup time(%) Baseline xx/xx (%) xx/xx (%) Days 1-183 xx/xx (%) xx/xx (%)

Note: Lesion rate (days) is defined as number of days with lesions divided by the number of days in the observation period.

Note: The overall rate is presented where numerator and denominator are summed across subjects.

Program: Date Produced: mm/dd/yy

Programming Notes:

- Present results for Baseline and Days 1-183.
- A day with lesions is a day for which LESIONS='Yes'.
- Number this table 14.2.2.1 and produce a similar table (14.2.2.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.2.3.1: Descriptive Summary of Individual Subject Lesion Rates by Treatment Group and Observation Period mTTT Population

| mITT Popula | ation | |
|-------------------------------------|----------------|------------|
| Visit | | |
| Statistic | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| Baseline | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Total subjects w/ at least 1 day of | n (%) | n (%) |
| lesions | | |
| D 1 102 | | |
| Days 1-183 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Total subjects w/ at least 1 day of | n (%) | n (%) |
| lesions | | |
| Change from Baseline (Days 1-183) | | |
| n | XX | XX |
| Mean | XX.XX | xx.xx |
| SD | XX.XXX | XX.XXX |
| Median | XX.XX | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| P-Value (vs. Placebo)[1] | 0.xxxx | |

Note: Lesion rate (days) is defined as number of days with lesions divided by the number of days in the observation

[1]P-value based on Wilcoxon rank sum test.

Programming Notes:

Program: Date Produced: mm/dd/yy

- Present results for Baseline and Days 1-183.
- A day with lesions is a day for which LESIONS='Yes'.
- $\bullet$  Number this table 14.2.3.1 and produce a similar table (14.2.3.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.2.4.1: Frequency of Recurrences at 6 Months After Maintenance Dose by Treatment Group mITT Population

| | GEN-003 60 ug/ | | P-value[1] |
|-----------------------------------|----------------|---------|------------|
| Statistic | M2 50 ug | Placebo | |
| | N=xx | N=xx | |
| Number of Recurrences at 6 Months | | | |
| after Maintenance Dose | | | 0.xxxx |
| n | XX | XX | |
| Mean | XX.XX | xx.xx | |
| SD | xx.xxx | XX.XXX | |
| Median | XX.XX | XX.XX | |
| | xx.x, xx.x | xx.x, | |
| Min, Max | | XX.X | |

Note: Recurrences refer to subject-reported recurrences.

[1]P-value based on Wilcoxon rank sum test.

Program: Date Produced: mm/dd/yy

Programming Notes:

 $\bullet$  Number this table 14.2.4.1 and produce a similar table (14.2.4.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.2.5.1: Proportion of Subjects Who Are Recurrence Free at 6 Months After Maintenance Dose

mITT Population Variable P-value[1] GEN-003 60 ug/ Statistic M2 50 ug Placebo N=xxN=xxRecurrence Free at 6 Months after Maintenance Dose\* 0.xxxx Yes n (%) n (%) n (%) No n (%) Unknown n (%) n (%)

[1] From a chi-square test of homogeneity of proportions (excluding Unknown counts).

Program: Date Produced: mm/dd/yy

Programming Notes:

• Number this table 14.2.5.1 and produce a similar table (14.2.5.2) for the PP population

<sup>\* &#</sup>x27;Yes' includes subjects who do not have a recurrence from Maintenance Dose through 6 months after Maintenance Dose.
'No' includes subjects who do have a recurrence from Maintenance Dose through 6 months after Maintenance Dose.
'Unknown' includes subjects who discontinue prior to 6 months after Maintenance Dose and have not had a recurrence prior to discontinuation.

Protocol: [Protocol number] page x of y

Table 14.2.6.1: Time to First Recurrence After Maintenance Dose  $$\tt mITT$$  Population

| Statistic | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
|---|---|---|
| Number with recurrence (%) | xx (xx.x) | xx (xx.x) |
| Number Censored (%) | xx(xx.x) | xx(xx.x) |
| Time to first | | |
| recurrence* | | |
| 25 <sup>th</sup> Percentile (95% CI) | xx(xx.x,xx.x) | xx(xx.x,xx.x) |
| Median (95% CI) | xx(xx.x,xx.x) | xx(xx.x,xx.x) |
| 75 <sup>th</sup> Percentile (95% CI) | xx(xx.x,NE) | xx(xx.x,NE) |
| Min, Max | xx,xx | xx,xx |
| K-M Estimate[1] (95% | | |
| CI) | x.xxx(x.xxx,x.xxx) | x.xxx(x.xxx,x.xxx) |
| Log rank test | 0.xxxx | |
| vs. Placebo p-value | | |

<sup>\*</sup> The number of days from Maintenance Dose to the day the subject experienced a recurrence, or the censoring day that the subject was last known to be recurrence-free. NE = Not Estimable CI = Confidence Interval K-M = Kaplan-Meier

[1] Percent of event-free subjects

Program: Date Produced: mm/dd/yy

#### Programming Notes:

• Number this table 14.2.6.1 and produce a similar table (14.2.6.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.2.7.1: Descriptive Summary and Analysis of Mean Lesion Outbreak Duration Over 6 Months After Maintenance Dose

| 11111 | i ropulacion | | |
|-------------------------------------|----------------|------------|---------|
| Visit | | | |
| Statistic | GEN-003 60 ug/ | | P-value |
| | M2 50 ug | Placebo | [1] |
| | N=xx | | |
| 6 Months After Maintenance Dose | | | 0.xxxx |
| n | XX | XX | |
| Mean | XX.XX | XX.XX | |
| SD | XX.XXX | XX.XXX | |
| Median | XX.XX | XX.XX | |
| Min, Max | XX.X, XX.X | XX.X, XX.X | |
| Total subjects w/ at least 1 day of | n (%) | n (%) | |
| lesions | | | |

Note: Mean lesion outbreak duration is defined for each subject as the average number of days with lesions per outbreak (recurrence) during the period of interest. Subjects with no recurrences during the period of interest are excluded from the analysis.

[1]P-value based on Wilcoxon rank sum test.

Program: Date Produced: mm/dd/yy

Programming Notes:

- A day with lesions is a day for which LESIONS='Yes'.
- Number this table 14.2.7.1 and produce a similar table (14.2.7.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.2.8.1: Summary of Antiviral Medication Use After Maintenance Dose

| mITT Population | | |
|---|---|---|
| Variable | | |
| Statistic | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
| Antiviral Medication Use After | | |
| Maintenance Dose | | |
| Yes | n (응) | n (%) |
| No | n (%) | n (%) |

Program: Date Produced: mm/dd/yy

Programming Notes:

• Antiviral medications are defined as medications with an ATC2 Class of 'ANTIVIRALS FOR SYSTEMIC USE'

 $\bullet$  Number this table 14.2.8.1 and produce a similar table (14.2.8.2) for the PP population

Protocol: [Protocol number] page x of y

Table 14.3.1.1: Frequency Table of All Adverse Events by SOC, Preferred Term, and Treatment

Safety Population

| Safety Population | | |
|---------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With AEs | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |

Note: Adverse event mapping was based on the MedDRA Version xx.x thesaurus.

Note: Subjects who have the same event more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Protocol: [Protocol number] page x of y

Table 14.3.1.2: Frequency Table of All Adverse Events by SOC, Preferred Term, Treatment, and Severity

Safety Population Severity: Grade 1 (Mild)

| peverity. Grad | ac = (111±±a) | |
|---------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With AEs | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |


Note: Subjects who have the same event more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Programming Note: Produce a subtable for each level of severity (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-threatening).

Protocol: [Protocol number] page x of y

Table 14.3.1.3: Frequency Table of All Adverse Events by SOC, Preferred Term, Treatment, and Causality

Safety Population

Relationship to Investigational Product: Likely

| | GEN-003 60 ug/ | |
|---------------------|----------------|---------|
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| 110101100 101 | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With AEs | (/ | (, |
| 1200 | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |


Note: Subjects who have the same event more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Programming Note: Produce a subtable for each level of causality/relationship to vaccine (Likely, Unlikely).
Protocol: [Protocol number] page x of y

Table 14.3.1.4: Frequency Table of All Adverse Events Leading to Discontinuation of Dosing by SOC, Preferred Term and Treatment

Safety Population

| salety rop | Jaracron | |
|---------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With AEs | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |


Note: Subjects who have the same event more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Protocol: [Protocol number] page x of y

Table 14.3.1.5: Frequency Table of Subjects with Adverse Events of Special Interest by SOC, Preferred Term and Treatment

Safety Population

| | Paracron | |
|---------------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With an Adverse | | |
| Event of Special Interest | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| 1 | | |


Note: Subjects who have the same event of Special Interest more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event of Special Interest within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Protocol: [Protocol number] page x of y

Table 14.3.1.6: Frequency Table of All Adverse Events with ≥ 5% Occurrence by SOC, Preferred Term, and Treatment

| Safety Population | | |
|---------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With AEs | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |


Note: Subjects who have the same event more than once are counted only once for the Preferred Term. Subjects who have more than one adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

### Programming Notes:

• Include all SOC/PT where the active treatment group has a ≥ 5% occurrence rate for that SOC/PT.

Protocol: [Protocol number] page x of y

Table 14.3.1.7: Summary of Local Reactions and Systemic Events Occurring Within 7 Days Postdose by Treatment and Maximum Severity

Safety Population

| | | GEN-003 60 ug/ | |
|-----------------------------------------|-------|----------------|----------|
| Local Reactions and | Grade | M2 50 ug | Placebo |
| Systemic Events | [1] | N=xx | N=xx |
| Any Local Reaction | Any | n (x.x%) | n (x.x%) |
| or Systemic Event | 1 | n (x.x%) | n (x.x%) |
| or systemic Event | 2 | | 4 0.1 |
| | 3 | | 4 0.1 |
| | 4 | | |
| | 4 | n (x.x%) | n (x.x%) |
| 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | - | ( 0 ) | 4 0) |
| Any Local Reaction | Any | n (x.x%) | n (x.x%) |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| Pain | Any | n (x.x%) | n (x.x%) |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| Tenderness | Any | n (x.x%) | n (x.x%) |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| Swelling | Any | n (x.x%) | n (x.x%) |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| | | , , | , , |
| Swelling (mm) | Any | n (x.x%) | n (x.x%) |

| | | GEN-003 60 ug/ | |
|---------------------|----------|----------------|----------|
| I and Deschions and | Consider | - | Dlasalas |
| Local Reactions and | Grade | M2 50 ug | Placebo |
| Systemic Events | [1] | N=xx | N=xx |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| | Any | n (x.x%) | n (x.x%) |
| | 1 | n (x.x%) | n (x.x%) |
| | 2 | n (x.x%) | n (x.x%) |
| | 3 | n (x.x%) | n (x.x%) |
| | 4 | n (x.x%) | n (x.x%) |
| Redness (mm) | | | |
| Any Systemic Event | ETC | n (x.x%) | n (x.x%) |
| Fever | ETC | n (x.x%) | n (x.x%) |
| Headache | ETC | n (x.x%) | n (x.x%) |
| Chills | ETC | n (x.x%) | n (x.x%) |
| Fatigue | ETC | n (x.x%) | n (x.x%) |
| Nausea | ETC | n (x.x%) | n (x.x%) |
| Diarrhea | ETC | n (x.x%) | n (x.x%) |
| Vomiting | ETC | n (x.x%) | n (x.x%) |
| Muscle aches | ETC | n (x.x%) | n (x.x%) |
| | | , , | . , |
| Any Local Reaction | | n (x.x%) | n (x.x%) |
| or Systemic Event | | | , |
| Any Local Reaction | | n (x.x%) | n (x.x%) |
| Pain | | n (x.x%) | n (x.x%) |
| ETC | | | |
| | | | l . |

Program: Date Produced: mm/dd/yy

- Information comes from the Diary Card
- If a subject has multiple of the same events, take the maximum severity.
- During the 7 day period after the (Days 1-7) a subject should only be counted one time. If a subject has a sign/symptom at least once during that 7 day interval the subject is counted for that sign/symptom.
- Watch page breaks. Please try and keep all the grades together for a sign/symptom.
- Do not include Grade=0 as Grades of 0 imply "None" or no event.
- Fever is based on Temperature (F) which is collected on the Diary Card. See Appendix 2 in the protocol for grade definitions. Grade 1 = 100.4-101.1; Grade 2 = 101.2-102.0; Grade 3 = 102.1-104; Grade 4 > 104.

• For Redness (mm) and Swelling (mm), see also Appendix 2 in the protocol. For both redness and swelling: Grade 1 = 2.5-5 cm; Grade 2 = 5.1-10 cm; Grade 3 = >10cm; Grade 4 is Necrosis or exfoliative dermatitis, which we won't be able to determine and will be handled separately as an AE.

Protocol: [Protocol number] page x of y

Table 14.3.1.8: Descriptive Summary of Duration (days) of Systemic Events and Local Reactions by Treatment

Safety Population

| | | | Sai |
|------------------------|------------|----------------|---------|
| Systemic<br>Events and | | GEN-003 60 ug/ | |
| Local | | M2 50 ug | Placebo |
| Reactions | Statistic | N=xx | N=xx |
| Fever | N | XX | XX |
| | Median | XX.X | XX.X |
| | Minimum | XX | XX |
| | Maximum | XX | XX |
| Headache | N | XX | XX |
| | Median | XX.X | XX.X |
| | Minimum | XX | XX |
| | Maximum | XX | XX |
| Chills | N | | |
| CHILLS | Median | XX | XX |
| | Minimum | XX.X | XX.X |
| | Maximum | XX | XX |
| | Maxillulli | XX | XX |
| Fatigue | N | XX | XX |
| | Median | XX.X | XX.X |
| | Minimum | XX | XX |
| | Maximum | XX | XX |
| Nausea | N | XX | XX |
| | Median | XX.X | XX.X |
| | Minimum | XX | XX |
| | Maximum | XX | XX |
| Dairrhea | N | | |
| Dallinea | Median | | |
| ETC | ETC | | |
| Drogram. | | | |

Program: Date Produced: mm/dd/yy

Programming Notes:

• Information comes from the Diary Card

• For start date, use the date from when the symptom is first recorded on the card (severity >0). For the stop date, use the date when the symptom is last present on the card (severity > 0). If a stop date is not available, then this needs to be given to the CDM.

Protocol: [Protocol number] page x of y

Table 14.3.1.9: Summary of Antipyretic/Analgesic Medications Taken Within 7 Days after Maintenance Dose by Treatment Group, Drug Class and Preferred Term

Safety Population

| Preferred Term | GEN-003 60 ug/<br>M2 50 ug<br>N=xx | Placebo<br>N=xx |
|---|---|---|
| Any Anti-Fever/Anti-Pain Medication | n (x.x%) | n (x.x%) |
| Preferred Term 1 | n (x.x%) | n (x.x%) |
| Preferred Term 2 | n (x.x%) | n (x.x%) |
| Preferred Term 3 | n (x.x%) | n (x.x%) |
| etc. | | |

Program: Date Produced: mm/dd/yy

## Programming Note:

• Antipyretic/analgesic medications are defined as medications with an ATC2 Class of 'ANALGESICS' or 'ANTIINFLAMMATORY AND ANTIRHEUMATIC PRODUCTS'

Protocol: [Protocol number] page x of y

Table 14.3.2.1: Frequency Table of Subjects with Serious Adverse Events by SOC, Preferred Term and Treatment
Safety Population

| Salety Population | |
|---|---|
| GEN-003 60 ug/ | |
| M2 50 ug | Placebo |
| N=xx | N=xx |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| x (x.x) | x (x.x) |
| | X (X.X) |


Note: Subjects who have the same serious adverse event more than once are counted only once for the Preferred Term. Subjects who have more than one serious adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

Protocol: [Protocol number] page x of y

Table 14.3.2.2: Frequency Table of Subjects with Medically Attended Adverse Events by SOC, Preferred Term and Treatment

| Safety Population | | |
|---------------------------|----------------|---------|
| | GEN-003 60 ug/ | |
| | M2 50 ug | Placebo |
| | N=xx | N=xx |
| MedDRA SOC | | |
| Preferred Term | | |
| Total Number (%) of | x (x.x) | x (x.x) |
| Subjects With a Medically | | |
| Attended AE | | |
| SOC1 | x (x.x) | x (x.x) |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOC2 | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |
| SOCn | | |
| PT1 | x (x.x) | x (x.x) |
| PT2 | x (x.x) | x (x.x) |


Note: Subjects who have the same medically attended adverse event more than once are counted only once for the Preferred Term. Subjects who have more than one medically attended adverse event within a System Organ Class are counted only once in that System Organ Class.

Program: Date Produced: mm/dd/yy

**List of Statistical Listings for GEN-003-005** 

| Listing No. | Listing Title | Analysis<br>Population |
|---|---|---|
| 16.2.1 | Subject Disposition and Reasons for Discontinuation From Study | Safety |
| 16.2.2.1 | Protocol Deviations by Subject | Safety |
| 16.2.2.2 | Randomization and Analysis Populations by Subject | Safety |
| 16.2.3 | Subjects Excluded from the Per Protocol Analysis Population | Safety |
| 16.2.4.1 | Baseline Demographics by Subject | Safety |
| 16.2.4.2 | Medical History by Subject | Safety |
| 16.2.4.3 | Prior Medications by Subject | Safety |
| 16.2.4.4 | Concomitant Medications by Subject | Safety |
| 16.2.5.1 | Dosing Status by Subject | Safety |
| 16.2.5.2 | Dosing Date/Time by Subject | Safety |
| 16.2.6.1 | Electronic Diary Data by Subject | Safety |
| 16.2.6.2 | EQ-5D-5L Data by Subject | Safety |
| 16.2.7.1 | Systemic Events (Diary Card) by Subject | Safety |
| 16.2.7.2 | Local Reactions (Diary Card) by Subject | Safety |
| 16.2.7.3 | Adverse Events by Subject | Safety |
| 16.2.7.4 | Serious Adverse Events by Subject | Safety |
| 16.2.7.5 | Adverse Events Associated with Discontinuation of Dosing by Subject | Safety |
| 16.2.7.6 | Adverse Events Leading to Death by Subject | Safety |
| 16.2.7.7 | Medically Attended Adverse Events by Subject | Safety |
| 16.2.7.8 | Adverse Events of Special Interest by Subject | Safety |
| 16.2.8.1 | Heina Pragnanay Tagt Pagulta by Subject | Safety |
| 16.2.8.2 | Urine Pregnancy Test Results by Subject Pregnancy Results by Subject | Safety |
| 10.4.0.4 | rregnancy results by Subject | Salety |

Protocol: [Protocol number] page x of y

Listing 16.2.1: Subject Disposition and Reasons for Discontinuation From Study

Safety Population

| | | Safety Po | <del>-</del> | T | |
|---|---|---|---|---|---|
| Treatment | Subject | Subject | Disposition | Reason(s) for | Discontinuation |
| | Number | Status | Date | Discontinuation | Explanation |
| GEN-003 60 ug / M2 50 ug | XXXX | | ddmmmyyyy | Completed | |
| | XXXX | | | Withdrew consent | |
| | | | | due to AE | |
| | XXXX | | | Withdrew consent | |
| | | | | not due to AE | |
| | XXXX | | | Lost to Follow-up | |
| | | | | Non-compliance | |
| Placebo | XXXX | | | Investigator | |
| | | | | discretion | |
| | XXXX | | | Sponsor request | |
| | XXXX | | | Death | |
| | XXXX | | | Site termination | |
| | XXXX | | | Study termination | |
| | XXXX | | | | |

Program: Date Produced: mm/dd/yy

- "Subject Status": If DSDECOD = "Subject completed" then "Subject Status" = "Completed study". If DSDECOD is ≠ "Subject completed" then "Subject Status" = "Did not complete study".
- Sort by treatment, subject number.

Protocol: [Protocol number] page x of y

# Listing 16.2.2.1: Protocol Deviations by Subject

Safety Population

| Subject | Deviations | Deviation Type | Deviation Type | Description of | Site |
|---|---|---|---|---|---|
| Number | Date | - Subject | - Site | Deviation | Corrective |
| | | | | | Action |
| XXXX | ddmmmyyyy | Subject did not meet | Missed | | |
| | | eligibility criteria | procedure | | |
| | ddmmmyyyy | Subject received wrong | Out of window | | |
| | | treatment or incorrect | procedure | | |
| | | dose | | | |
| | ddmmmyyyy | Subject received | Consent | | |
| | | prohibited concomitant | process error | | |
| | | medication | | | |
| | | Subject received a vaccine | Noncompliance | | |
| | | in excluded time period | | | |
| | | Subject used suppressive | Other | | |
| | | antiviral therapy | | | |
| XXXX | | Consent process error | | | |
| XXXX | | Noncompliance | | | |
| XXXX | | Other | | | |
| XXXX | | | | | |
| XXXX | | | | | |
| XXXX | | | | | |
| XXXX | | | | | |
| XXXX | | | | | |
| | xxxx xxxx xxxx xxxx xxxx xxxx xxxx | Number Date xxxx ddmmmyyyy ddmmmyyyy ddmmmyyyy xxxx xxxx xxxx xxxx xxxx xxxx xxxx | Number Date - Subject xxxx ddmmmyyyy Subject did not meet eligibility criteria ddmmmyyyy Subject received wrong treatment or incorrect dose ddmmmyyyy Subject received prohibited concomitant medication Subject received a vaccine in excluded time period Subject used suppressive antiviral therapy xxxx Consent process error xxxx Noncompliance xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xx | Number Date - Subject - Site xxxx ddmmmyyyy Subject did not meet eligibility criteria procedure ddmmmyyyy Subject received wrong treatment or incorrect dose ddmmmyyyy Subject received procedure dose Consent process error Subject received a vaccine in excluded time period Subject used suppressive antiviral therapy xxxx Consent process error xxxx Noncompliance xxxx Other xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xx | Number Date - Subject - Site Deviation xxxx ddmmmyyyy Subject did not meet eligibility criteria procedure ddmmmyyyy Subject received wrong treatment or incorrect dose ddmmmyyyy Subject received prohibited concomitant medication Subject received a vaccine in excluded time period Subject used suppressive antiviral therapy xxxx Consent process error xxxx Noncompliance xxxx Other xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xxxx Xx |

Program: Date Produced: mm/dd/yy

- Deviation information will come from the Protocol Deviations CRF.
- Sort by treatment, subject number, and deviations date.

Protocol: [Protocol number] page x of y

# Listing 16.2.2.2: Randomization and Analysis Populations by Subject

Safety Population

| Treatment | Subject | Informed | Randomization | Did Subject Meet | If no, | mITT | Safety | Per |
|---|---|---|---|---|---|---|---|---|
| | Number | Consent | Date | all of the | Criteria | Population | Population | Protocol |
| | | Date | | Eligibility | Not Met | | | Population |
| | | | | Criteria | | | | |
| GEN-003 60 | XXXX | ddmmmyyyy | ddmmmyyyy | Yes | | Yes | Yes | Yes |
| ug / M2 50 | | | | | | | | |
| ug | | | | | | | | |
| | XXXX | | | No | | No | No | No |
| | XXXX | | | | | | | |
| Placebo | XXXX | | | | | | | |
| | XXXX | | | | | | | |
| | XXXX | | | | | | | |
| | XXXX | | | | | | | |
| | XXXX | | | | | | | |
| | | • | | | | | | |

Program: Date Produced: mm/dd/yy

- Sort by treatment, subject number.
- Information comes from Randomization and Eligibility-Demographics CRFs.

Protocol: [Protocol number] page x of y

Listing 16.2.3: Subjects Excluded from the Per Protocol Analysis Population

Safety Population

| Treatment | Subject | Reason for Exclusion from |
|--------------------------|---------|--------------------------------------|
| | Number | Per Protocol Population |
| GEN-003 60 ug / M2 50 ug | XXXX | Inclusion/exclusion criteria not met |
| | XXXX | Daily electronic diary noncompliance |
| | XXXX | Had an important protocol deviation |
| Placebo | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |
| | XXXX | |

Program: Date Produced: mm/dd/yy

- More than one reason may be listed for a subject.
- Sort by treatment and subject number.

Protocol: [Protocol number] page x of y

Listing 16.2.4.1: Baseline Demographics by Subject

Safety Population

| | | | | ecy ropuración | | |
|---|---|---|---|---|---|---|
| Treatment | Subject | Age | Sex | Ethnicity | Race | Weight |
| | Number | | | | | (lbs) |
| GEN-003 60 ug / | XXXX | | | Hispanic | White | |
| M2 50 ug | | | | | | |
| | XXXX | | | Non-Hispanic | Black or African | |
| | | | | | American | |
| | XXXX | | | | Asian | |
| | XXXX | | | | American Indian or | |
| | | | | | Alaska Native | |
| | XXXX | | | | Native Hawaiian or | |
| | | | | | Other Pacific Islander | |
| Placebo | XXXX | | | | Other, specify | |
| | XXXX | | | | | |
| | XXXX | | | | | |

Program: Date Produced: mm/dd/yy

- Data comes from the Eligibility-Demographics CRF.
- Sort by treatment, subject number.

Protocol: [Protocol number] page x of y

## Listing 16.2.4.2: Medical History by Subject

Safety Population

| Treatment | Subject Number | SOC | Preferred | Term | Verbatim | Status |
|---|---|---|---|---|---|---|
| GEN-003 60 ug / M2 50 ug | XXXX | | | | | Ongoing |
| | XXXX | | | | | Intermittent |
| | XXXX | | | | | Resolved |
| Placebo | XXXX | | | | | |
| | XXXX | | | | | |
| | XXXX | | | | | |
| | | | | • | | |

Program: Date Produced: mm/dd/yy

# Programming Notes:

• Sort by treatment, subject number, SOC and Preferred Term.

Protocol: [Protocol number] page x of y

## Listing 16.2.4.3: Prior Medications by Subject

Safety Population

| Treatment | Subject | ATC Text Level 2/ | Route | Start Date | Stop Date | Ongoing |
|---|---|---|---|---|---|---|
| | Number | Preferred Name/ | | | - | |
| | | Medication | | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| GEN-003 60 ug / M2 50 ug | XXXX | mmmmmmmmmmmmm | Oral | ddmmmyyyy | ddmmmyyyy | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Topical | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Subcutaneous | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppp/ | | | | |
| | | mmmmmmmmmmmmm | Transdermal | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppp/ | | | | |
| Placebo | XXXX | mmmmmmmmmmmmm | Intraocular | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Intramuscular | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Inhalation | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | | mmmmmmmmmmmmm | Intraperitoneal | | | |
| | | • • • | Nasal | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Vaginal | | | |

Program:

Date Produced: mm/dd/yy

- Sort by treatment, subject, start date, stop date, and medication.
- Prior meds are any meds with a start date BEFORE date of maintenance dose (Day 1).
- Prior Meds will be coded.
- Please try to keep subject data together. Depending on number of con meds per subject, this may not be possible.

Protocol: [Protocol number] page x of y

# Listing 16.2.4.4: Concomitant Medications by Subject

Safety Population

| Treatment | Subject | ATC Text Level 2/ | Route | Start Date | Stop Date | Ongoing |
|---|---|---|---|---|---|---|
| | Number | Preferred Name/ | | | - | |
| | | Medication | | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| GEN-003 60 ug / M2 50 ug | XXXX | mmmmmmmmmmmmm | Oral | ddmmmyyyy | ddmmmyyyy | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Topical | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmmm | Subcutaneous | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | | mmmmmmmmmmmmm | Transdermal | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| Placebo | XXXX | mmmmmmmmmmmmm | Intraocular | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Ppppppppppppppppppp/ | | | | |
| | XXXX | mmmmmmmmmmmm | Intramuscular | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppppppppppppppppppppppp | | | | |
| | XXXX | mmmmmmmmmmm | Inhalation | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppppppppppppppppppppppp | | | | |
| | | mmmmmmmmmmmmm | Intraperitoneal | | | |
| | | | Nasal | | | |
| | | Xxxxxxxxxxxx/ | | | | |
| | | Pppppppppppppppppppppppppppppppppppppp | | | | |
| | XXXX | mmmmmmmmmmmmm | Vaginal | | | |

Program:

Programming Notes:

Date Produced: mm/dd/yy

- Sort by treatment, subject, start date, stop date, and medication.
- Concomitant meds are any meds which started on or after the date of maintenance dose (Day 1), or which started before date of maintenance dose and continued beyond date of maintenance dose.
- Concomitant Meds will be coded.
- Please try to keep subject data together. Depending on number of con meds per subject, this may not be possible.

Protocol: [Protocol number] page x of y

# Listing 16.2.5.1: Dosing Status by Subject

| barcey roparación | | | |
|---|---|---|---|
| Treatment | Subject<br>Number | Was Dose Temporarily Delayed? | Reason for<br>Temporary Delay |
| GEN-003 60 ug / M2<br>50 ug | xxxx | Yes | Fever |
| | | No | Other acute<br>illness |
| Placebo | xxxx | | |

Program: Date Produced: mm/dd/yy

- Sort by treatment, subject.
- Data collected on Study Drug Discontinuation CRF.

Protocol: [Protocol number] page x of y

# Listing 16.2.5.2: Dosing Date/Time by Subject

Safety Population

| | Salety Population | | | |
|---|---|---|---|---|
| Treatment | Subject Number | Dose Date | Dose Time | Location |
| GEN-003 60 ug / M2 50 ug | XXXX | ddmmmyyyy | hh:mm | Left deltoid |
| | | | | Right deltoid |
| | xxxx | ddmmmyyyy | hh:mm | |
| Placebo | XXXX | ddmmmyyyy | hh:mm | |
| | XXXX | ddmmmyyyy | hh:mm | |
| 1 | | I | l | [ |

Program: Date Produced: mm/dd/yy

- Sort by treatment, subject.
- Data collected on Study Immunization CRF.

Protocol: [Protocol number] page x of y

# Listing 16.2.6.1: Electronic Diary Data by Subject

Safety Population

| Treatment | Subject | Date | Lesions | # | Open | Prodrome | Itching | Pain | Pain | Draining | Swelling |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Number | | | Lesions | Lesion | | Score | Score | During | or | Score |
| | | | | | | | | | Urination | Discharge | |
| | | | | | | | | | Score | Score | |
| GEN-003 | XXXX | ddmmmyyyy | Yes | XX | Yes | Yes | Х | Х | X | X | Х |
| 60 ug / | 212121 | admining y y y | 105 | 2222 | 105 | 105 | 25 | 21 | 21 | 21 | 21 |
| M2 50 ug | | | | | | | | | | | |
| M2 30 ug | | | No | | No | No | | | | | |
| | | | NO | | NO | No | | | | | |
| Placebo | xxxx | | | | | | | | | | |
| | XXXX | | | | | | | | | | |

Program: Date Produced: mm/dd/yy

- Sort by treatment, subject, date.
- Data comes from Signs and Symptoms diary.

Protocol: [Protocol number] page x of y

# Listing 16.2.6.2: EQ-5D-5L Data by Subject

Safety Population

| Treatment | Subject | Date | Mobility | Self-Care | Usual | Pain/ | Anxiety/Depression | Health |
|---|---|---|---|---|---|---|---|---|
| 11000 | Number | 2430 | 110211101 | 3011 3013 | Activities | Discomfort | Immicos, sopiessiem | Rating |
| GEN-003 | XXXX | ddmmmyyyy | No | No | No | No pain | Not anxious | XX |
| 60 ug / | | | problems | problems | problems | I I I I I I I I I I I I I I I I I I I | | |
| M2 50 ug | | | 1 | F-000-00000 | F = 0.0 = 00 | | | |
| 5 | | | Slight | Slight | Slight | Slight | Slightly anxious | |
| | | | problems | problems | problems | pain | | |
| | | | Moderate | Moderate | Moderate | Moderate | Moderately anxious | |
| | | | problems | problems | problems | pain | _ | |
| | | | Severe | Severe | Severe | Severe | Severely anxious | |
| | | | problems | problems | problems | pain | _ | |
| | | | Unable | Unable to | Unable to | Extreme | Extremely anxious | |
| | | | to walk | wash/dress | do usual | pain | _ | |
| | | | | | activities | | | |
| Placebo | XXXX | | | | | | | |
| | XXXX | | | | | | | |

Program:

Date Produced: mm/dd/yy

- Sort by treatment, subject, date.
- Data comes from EQ-5D-5L CRF.

Protocol: [Protocol number] page x of y

Listing 16.2.7.1: Systemic Events (Diary Card) by Subject

Safety Population Visit Temperature Chills Fatigue Nausea Treatment Subject Date Headache Etc. Number (F) GEN-003 60 ug / M2 50 ug XXXX Day 1 Pre ddmmmyyyy XX.X 0 0 Day 1 (1hr) 1 1 1 Day 1 Day 2 3 3 3 3 Day 3 Day 4 Dav 5 Day 6 Day 7 Placebo XXXX

Date Produced: mm/dd/yy

Grade 0 = None; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe Program:

- Sort by treatment, subject, and visit.
- Data comes from Body Symptoms-Reactions Log CRF; for visit and time information, use the variable DCNOMDAT.
- Diary Cards are filled out for the 7 days following the maintenance dose.
- Page break by subject.
- Always include the first 7 days after the maintenance dose; if additional days are captured and the symptoms are all = 0 (None), then do not present on listing.

Protocol: [Protocol number] page x of y

Listing 16.2.7.2: Local Reactions (Diary Card) by Subject

Safety Population

| Treatment | Subject Number | | Date | Pain | Tenderness | Swelling | Swelling (mm) | Redness (mm) |
|---|---|---|---|---|---|---|---|---|
| GEN-003 60 ug / M2 50 ug | XXXX | Day 1 Pre | ddmmmyyyy | 0 | 0 | 0 | XXX | XXX |
| | | Day 1 (1hr) | | 1 | 1 | 1 | | |
| | | Day 1 | | 2 | 2 | 2 | | |
| | | Day 2 | | 3 | 3 | 3 | | |
| | | Day 3 | | | | | | |
| | | Day 4 | | | | | | |
| | | Day 5 | | | | | | |
| | | Day 6 | | | | | | |
| | | Day 7 | | | | | | |
| Placebo | XXXX | | | | | | | |

Date Produced: mm/dd/yy

Grade 0 = None; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe

Program:

- Sort by treatment, subject, and visit.
- Diary Cards are filled out for the 7 days following the maintenance dose.
- Data comes from Body Symptoms-Reactions Log CRF; for visit and time information, use the variable DCNOMDAT.
- Page break by subject.
- Always include the first 7 days after the maintenance dose; if additional days are captured and the symptoms are all = 0 (None), then do not present on listing.

Protocol: [Protocol number] page x of y

### Listing 16.2.7.3: Adverse Events by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject<br>Number | MedDRA SOC/<br>Preferred | Start<br>Date/ | Stop<br>Date/ | Severity [1] | Outcome | Action<br>Taken | AE<br>Related | Serious | AESI | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|
| | Term/ AE Verbatim | Day | Day | | | with<br>Study | To Study<br>Drug | | | |
| xx-xxx | | ddmmmyyyy<br>/<br>xxx | ddmmmyyyy<br>/<br>xxx | 1 | Fatal | Drug<br>None | Likely | Not Serious | Yes | Yes |
| | | | | 2 | Not<br>recovered | Dose<br>delayed | Unlikely | Death | No | No |
| | | | | 3 | Recovered | Drug<br>withdrawn | | Life<br>Threatening | | |
| | | | | 4 | Recovered<br>w/<br>sequelae | | | Hospitaliza<br>tion | | |
| | | | | | | | | Significant<br>Disability | | |
| | | | | | | | | Congenital Anomaly or Birth Defect | | |
| | | | | | | | | Other<br>medically<br>important<br>event | | |
| | 7.1 | | | | 41.11 | | | | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program: Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

### Listing 16.2.7.4: Serious Adverse Events by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject | MedDRA | Start | Stop | Severity | Outcome | Action | AE | Serious | AESI | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | SOC/ | Date/ | Date/ | [1] | | Taken | Related | | | |
| | Preferred | Day | Day | | | with | To Study | | | |
| | Term/ | | _ | | | Study | Drug | | | |
| | AE | | | | | Drug | _ | | | |
| | Verbatim | | | | | | | | | |
| XX-XXX | | ddmmmyyyy/ | ddmmmyyyy/ | 1 | Fatal | None | Likely | Death | Yes | Yes |
| | | XXX | XXX | | | | | | | |
| | | | | 2 | Not | Dose | Unlikely | Life | No | No |
| | | | | | recovered | delayed | | Threatening | | |
| | | | | 3 | Recovered | Drug | | Hospitaliza | | |
| | | | | | | withdrawn | | tion | | |
| | | | | 4 | Recovered | | | Significant | | |
| | | | | | w/ | | | Disability | | |
| | | | | | sequelae | | | | | |
| | | | | | | | | Congenital | | |
| | | | | | | | | Anomaly or | | |
| | | | | | | | | Birth | | |
| | | | | | | | | Defect | | |
| | | | | | | | | Other | | |
| | | | | | | | | medically | | |
| | | | | | | | | important | | |
| | | | | | | | | event | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program: Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- List out all AEs EXCEPT where Serious = 'No'.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

### Listing 16.2.7.5: Adverse Events Associated with Discontinuation of Dosing by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject | MedDRA SOC/ | Start | Stop | Severity | Outcome | Action | AE | Serious | AESI | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Preferred | Date/ | Date/ | [1] | | Taken | Related | | | |
| | Term/ | Day | Day | | | with | To Study | | | |
| | AE Verbatim | | | | | Study | Drug | | | |
| | | | | | | Drug | | | | |
| XX-XXX | | ddmmmyyyy/ | ddmmmyyyy/ | 1 | Fatal | Drug | Likely | Not Serious | Yes | Yes |
| | | XXX | XXX | | | withdrawn | | | | |
| | | | | 2 | Not | | Unlikely | Death | No | No |
| | | | | | recovered | | | | | |
| | | | | 3 | Recovered | | | Life | | |
| | | | | | | | | Threatening | | |
| | | | | 4 | Recovered | | | Hospitaliza | | |
| | | | | | w/ | | | tion | | |
| | | | | | sequelae | | | | | |
| | | | | | | | | Significant | | |
| | | | | | | | | Disability | | |
| | | | | | | | | Congenital | | |
| | | | | | | | | Anomaly or | | |
| | | | | | | | | Birth | | |
| | | | | | | | | Defect | | |
| | | | | | | | | Other | | |
| | | | | | | | | medically | | |
| | | | | | | | | important | | |
| | | | | | | | | event | | |
| | 7.1 | | | | | | | | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program: Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- List out all AEs where Action Taken = Drug withdrawn.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

### Listing 16.2.7.6: Adverse Events Leading to Death by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject | MedDRA SOC/ | Start | Stop | Severity | Outcome | Action | AE | Serious | AESI | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Preferred | Date/ | Date/ | [1] | | Taken | Related | | | |
| | Term/ | Day | Day | | | with Study | To Study | | | |
| | AE Verbatim | | | | | Drug | Drug | | | |
| XX-XXX | | ddmmmyyyy/<br>xxx | ddmmmyyyy/<br>xxx | 1 | Fatal | None | Likely | Death | Yes | Yes |
| | | | | 2 | | Dose<br>delayed | Unlikely | | No | No |
| | | | | 3 | | Drug | | | | |
| | | | | | | withdrawn | | | | |
| | | | | 4 | | | | | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program: Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- List out all AEs where Outcome=Fatal OR Serious=Death.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

### Listing 16.2.7.7: Medically Attended Adverse Events by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject | MedDRA SOC/ | Start | Stop | Severit | Outcome | Action | AE | Serious | AESI | MAAE | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Preferred | Date/ | Date/ | y [1] | | Taken | Related | | | | Type |
| | Term/ | Day | Day | | | with Study | To Study | | | | |
| | AE Verbatim | | | | | Drug | Drug | | | | |
| xx-xxx | | ddmmmyyyy | ddmmmyyyy | 1 | Fatal | None | Likely | Not Serious | Yes | Yes | ER |
| | | / | / | | | | | | | | Visit |
| | | XXX | XXX | | | | | | | | |
| | | | | 2 | Not | Dose | Unlikely | Death | No | | Other |
| | | | | | recovered | delayed | | | | | visit |
| | | | | 3 | Recovered | Drug | | Life | | | |
| | | | | | | withdrawn | | Threatening | | | |
| | | | | 4 | Recovered | | | Hospitaliza | | | |
| | | | | | W/ | | | tion | | | |
| | | | | | sequelae | | | | | | |
| | | | | | | | | Significant | | | |
| | | | | | | | | Disability | | | |
| | | | | | | | | Congenital | | | |
| | | | | | | | | Anomaly or | | | |
| | | | | | | | | Birth | | | |
| | | | | | | | | Defect | | | |
| | | | | | | | | Other | | | |
| | | | | | | | | medically | | | |
| | | | | | | | | important | | | |
| | | | | | | | | event | | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program: Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- List out all AEs where MAAE=Yes.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

## Listing 16.2.7.8: Adverse Events of Special Interest by Subject

Safety Population

Treatment: GEN-003 60 ug / M2 50 ug

| Subject | MedDRA SOC/ | Start | Stop | Severit | Outcome | Action | AE | Serious | AESI | MAAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Preferred | Date/ | Date/ | у [1] | | Taken | Related | | | |
| | Term/ | Day | Day | _ | | with Study | To Study | | | |
| | AE Verbatim | | | | | Drug | Drug | | | |
| xx-xxx | | ddmmmyyyy | ddmmmyyyy | 1 | Fatal | None | Likely | Not Serious | Yes | Yes |
| | | / | / | | | | | | | |
| | | XXX | XXX | | | | | | | |
| | | | | 2 | Not | Dose | Unlikely | Death | | No |
| | | | | | recovered | delayed | | | | |
| | | | | 3 | Recovered | Drug | | Life | | |
| | | | | | | withdrawn | | Threatening | | |
| | | | | 4 | Recovered | | | Hospitaliza | | |
| | | | | | w/ | | | tion | | |
| | | | | | sequelae | | | | | |
| | | | | | | | | Significant | | |
| | | | | | | | | Disability | | |
| | | | | | | | | Congenital | | |
| | | | | | | | | Anomaly or | | |
| | | | | | | | | Birth | | |
| | | | | | | | | Defect | | |
| | | | | | | | | Other | | |
| | | | | | | | | medically | | |
| | | | | | | | | important | | |
| | | | | | | | | event | | |

Note: Adverse event coding was done using the MedDRA Version xx.x dictionary.

[1] Severity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially life-threatening

AESI = Adverse Event of Special Interest

MAAE = Medically Attended Adverse Event

Program:

Date Produced: mm/dd/yy

- Sort by Treatment, Subject number, start date, stop date, SOC, PT.
- If "Ongoing" is checked, then AE Stop Date should be missing. Put "Ongoing" in the Stop Date column.
- List out all AEs where AESI=Yes.
- May need to use an 8-point font for this listing

Protocol: [Protocol number] page x of y

Listing 16.2.8.1: Urine Pregnancy Test Results by Subject
Safety Population

| Saissi isharasish | | | |
|---|---|---|---|
| Treatment | Subject Number | Date | Results |
| GEN-003 60 ug / M2 50 ug | XXXX | ddmmmyyyy | Negative |
| | | | Positive |
| | | | Not done |
| Placebo | | | |

Program:

Date Produced: mm/dd/yy

Programming Note:

• Sort by Treatment, Subject number.

Protocol: [Protocol number] page x of y

# Listing 16.2.8.2: Pregnancy Results by Subject

Safety Population
Treatment: GEN-003 60 ug / M2 50 ug

| Subject | Date | Date of | Expected | Date of | Date of | Date of | Date of | Other | Pregnancy | Status | Describe | Compli- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | | Last | Date of | Ultrasound | Amniocentesis | Chorionic | MSAFP/ | | Outcome | | | cations |
| | | Menstrual | Delivery | | | Villus | Serum | | | | | |
| | | Period | | | | Sampling | Markers | | | | | |
| XXXX | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | | Unknown | Healthy | | Yes |
| | | | | | | | | | | Baby | | |
| | | | | | | | | | Full term | Sick | X | No |
| | | | | | | | | | | Baby | | |
| | | | | | | | | | | (describe) | | |
| | | | | | | | | | Premature | Stillbirth | | |
| | | | | | | | | | Birth | | | |
| | | | | | | | | | Spontaneous | Congenital | | |
| | | | | | | | | | Miscarriage | Anomaly/ | X | |
| | | | | | | | | | | Birth defect | | |
| | | | | | | | | | | (describe) | | |
| | | | | | | | | | Elective | Multiple | | |
| | | | | | | | | | termination | Births(#) | | |

Program: Date Produced: mm/dd/yy

Programming Note:

• Sort by Treatment, Subject number.